CLINICAL TRIAL: NCT06201026
Title: Effects of Individualized, Home-based, Mobile App-guided Training to Reduce Fatigue in Patients With Newly and Advanced Diagnosed Multiple Sclerosis: a Randomized Controlled Trial.
Brief Title: Effects of Individualized Training to Reduce Fatigue in Patients With Newly and Advanced Diagnosed Multiple Sclerosis
Acronym: MovelySEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23CH024; ANSM (Other: 2023-A00535-40)
Record Dates: First submitted 2023-12-12; First posted 2024-01-11 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Sclerosis; Fatigue
Keywords: Fatigue; Neuromuscular function; Muscle characteristics; Physical capacity
MeSH Terms: conditions — Sclerosis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional exercise group in newly diagnosed patients with MS (SEP-R-TEM) (Active Comparator): Newly diagnosed patients with MS who will be part of the group doing traditional exercises
  Interventions: Other: Traditional exercise
- Individualized exercise group in newly diagnosed patients with MS (SEP-R-IND) (Experimental): Newly diagnosed patients with MS who will be part of the group doing individualized exercises
  Interventions: Other: Individualized exercise
- Traditional exercise group in advanced diagnosed patients with MS (SEP-A-TEM) (Active Comparator): Advanced diagnosed patients with MS who will be part of the group doing traditional exercises
  Interventions: Other: Traditional exercise
- Individualized exercise group in advanced diagnosed patients with MS (SEP-A-IND) (Experimental): Advanced diagnosed patients with MS who will be part of the group doing individualized exercises.
  Interventions: Other: Individualized exercise

INTERVENTIONS:
Other: Traditional exercise — Patients will perform aerobic and resistance exercises that are consistent with the exercise guidelines for MS patients at home
  Arms: Traditional exercise group in advanced diagnosed patients with MS (SEP-A-TEM); Traditional exercise group in newly diagnosed patients with MS (SEP-R-TEM)
Other: Individualized exercise — Patients will performed a mobile-app guided program at home designed to address identified individual disabilities such as loss of muscle strength or cardiorespiratory deconditioning.
  Arms: Individualized exercise group in advanced diagnosed patients with MS (SEP-A-IND); Individualized exercise group in newly diagnosed patients with MS (SEP-R-IND)

SUMMARY:
Multiple sclerosis (MS) is a chronic autoimmune inflammatory disease of the central nervous system. It is characterized by complex and heterogeneous symptoms. Chronic fatigue is the most reported symptom in MS patients (80%). Current pharmacological treatments for MS patients reduce the number of relapses and their severity but do not improve symptoms such as fatigue. Physical activity is a therapy that helps reduce this fatigue, in addition to improving muscular and cardiorespiratory functions. However, the results are not optimal because MS patients remain less active than the general population. The improvement of the benefits of exercise therapy could therefore be based on three approaches: personalization of the training program, home practice and early initiation.

DETAILED DESCRIPTION:
The objective of this study will be to investigate the effects of individualized home-training, guided by a mobile application, to reduce fatigue in patients with newly (N) and advanced (A) diagnosed MS.

ELIGIBILITY:
Inclusion criteria

* Relapsing-remitting MS (RRMS) defined according to the criteria of McDonald
* MS diagnosed less than 2 years ago or whose first symptoms are estimated to be less than 5 years old OR MS diagnosed more than 2 years ago and whose first symptoms are estimated to be less than 5 years old
* With a high level of fatigue, corresponding to an FSS score > 4
* Expanded Disability Status Scale (EDSS) score < 4
* Medical Research Council (MRC) testing ≥ 4 in all leg muscles
* Ability to walk for 10 minutes without stopping (self-reported)
* Have a mobile phone with internet access
* Affiliated with or benefiting from a social security scheme
* Have freely given their written consent after being informed of the aim, the procedure and the potential risks involved

Exclusion criteria

* Spasticity or severe cerebellar ataxia in either leg.
* Abnormal range of movement of the toes and/or ankle
* Musculoskeletal injury that impairs pedalling
* Appearance of a multiple sclerosis attack in the 90 days preceding the study
* Recent adjustment of any medication or drug that may have an impact on fatigue: treatment of neuropathic pain: anti-epileptic and/or taking stimulants for fatigue (e.g. modafinil, amantadine, fampridine...)
* History of comorbid illness or conditions that would compromise the subject's safety during the study
* Participation at the same time in another medical intervention study or having participated in such a study in the 30 days prior to this study
* Pregnant and breast-feeding women
* Patients who are unable to understand the purpose of the study and the conditions under which it will be conducted, or who are unable to give their consent.
* Patients deprived of their liberty or under guardianship

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) | Week 15
  Change in the chronic fatigue score assessed using the FSS questionnaire before and after the training programme. From 1 to 7.
  The higher the score, the greater the fatigue

SECONDARY OUTCOMES:
cross sectional area (µm2) of type IIA fibers from the vastus lateralis muscle biopsies | Week 17
  ONLY FOR MS-N PATIENTS
Muscle enzymatic activity (UI) | Week 17
  ONLY FOR MS-N PATIENTS
  The enzymatic activity is measured for the following enzymes :
  * Phosphofructokinase (PFK)
  * lactate dehydrogenase (LDH)
  * citrate synthase (CS)
  * cyclo-oxygenase (COx)
  Enzymatic activity is measured in units international (UI) It indicates the rate of enzymatic reaction catalyzed by the enzyme, expressed in micromoles of substrate transformed (or product formed) per minute.
Maximal oxygen uptake (VO2max) (ml/min) | Week 15
  Cardiac stress test
Percentage of voluntary activation (%) | Week 16
  Voluntary Activation of the extensor muscles of the knee by peripheral nerve stimulation
C-reactive protein (CRP) (mg/l) | Week 15
  Blood sample
Maximal voluntary contraction (MVC) of the knee extensor muscle measurement | Week 16
  Maximal isometric force (maximal voluntary contraction, MVC) of the knee extensor muscle
Maximal voluntary contraction (MVC) of the hand grip measurement | Week 16
Balance test (s) | Week 16
  This test, performed in unipedal support, consists of asking the subject to hold the unipedal position for as long as possible, on the lower limb of his choice.
Quality of life questionnaire (SEP-59) | Week 15
  Scale from 0 (worst quality of life) to 100 (best quality of life)
Epworth score | Week 15
  From 0 to 24
  The higher the score, the greater the degree of drowsiness
Pittsburgh Sleep Quality Index (PSQI) | Week 15
  From 0 to 21 The higher the score, the worse the quality of sleep
Hospital Anxiety and Depression scale (HAD) | Week 15
  From 0 to 42 The higher the score, the greater the anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe CAMDESSANCHE, PHD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No